CLINICAL TRIAL: NCT02737995
Title: A Pilot Feasibility Study on Iron Stores and Skeletal Muscle Metabolism in Chronic Heart Failure
Brief Title: Iron Stores and Skeletal Muscle Metabolism in Chronic Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00396
Record Dates: First submitted 2016-04-08; First posted 2016-04-14 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Heart Failure
Keywords: Iron deficiency
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iron Replacement (Experimental)
  Interventions: Drug: Ferric carboxymaltose infusion

INTERVENTIONS:
Drug: Ferric carboxymaltose infusion — Subjects with functional iron deficiency determined by the results of iron biomarker results at Visit 2 will receive a single dose of intravenous ferric carboxymaltose . The dose of Injectafer will be calculated from a modified Ganzoni equation adapted from previous heart failure clinical trials The maximum dose of Injectafer will be 750 mg. The calculated dose of Injectafer will be diluted in normal saline solution (4 mg/ml) and administered via a volumetric pump administered over 30 minutes.

SUMMARY:
Iron deficiency may contribute to exercise intolerance by altering mitochondrial oxidative capacity in skeletal muscle. Functional iron deficiency is common in heart failure patients, but the relationship to exercise intolerance and mitochondrial oxidative capacity is unknown. This is a pilot study to determine the feasibility of the use of specialized 31P-MRS and MRI techniques for measurement of skeletal muscle bioenergetics in patients with heart failure with and without functional iron deficiency.

DETAILED DESCRIPTION:
This study will obtain pilot feasibility data to explore the relationship between blood biomarkers of functional iron deficiency and skeletal muscle mitochondrial oxidative capacity with 31P-magnetic resonance spectroscopy (MRS) and imaging in heart failure patients.

Twenty (20) subjects will be recruited from the clinical practice of the NYU Advanced Cardiac Therapeutics group at NYU Langone Medical Center.

Twenty (20) subjects will be recruited from the practice of the NYU Advanced Cardiac Therapeutics group at NYU Langone Medical Center. The study will require a maximum of four (4) visits over a period of five (5) weeks. Eligibility for Visits 2-4 will be determined by the screening criteria in Visit 1. It is anticipated that 50% of the screened subjects at Visit 1 will be eligible to participate in Visit 2. Eligibility for participation in Visits 3 and 4 will be determined by the results of the iron biomarkers obtained at Visit 2. We anticipate that 50% of the subjects at Visit 2 will be eligible to participate in Visits 3 and 4. Only subject with functional iron deficiency will participate in Visits 3 and 4. There is no clinical care component for this study.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* Age 21-80 years
* Chronic heart failure >3 months with NYHA Class I-III symptoms

Exclusion Criteria:

* Presence of implantable defibrillator, permanent pacemaker not designed for safe use in 3T MRI stud
* Metallic implant or implants that are deemed not suitable for MRI scan on 3T
* Aneurysm clips, cochlear implants, presence of shrapnel in strategic locations, and metal in the eye
* Known claustrophobia or any other history of intolerance of MRI procedure
* Treated diabetes mellitus or hemoglobin A1c (HbA1c) >6.5%
* Any hospitalization <60 days
* Myocardial infarction or stroke < 6 months
* Estimated glomerular filtration rate <30 ml/min
* Weight <50 or >120 kg
* Systolic blood pressure <90 mmHg or > 160 mmHg
* Heart rate <50 or >100 beats per minute
* Resting oxygen saturation on room air <92%
* Hemoglobin <11 g/dl
* Serum phosphate below normal range (<2.4 mg/dl)
* Liver function tests (AST, ALT, Alk Phos, or Total Bilirubin) >twice upper limit of normal range
* Pregnancy or current breastfeeding
* Exercise limitation primarily due to valvular heart disease, lung disease, neuromuscular disease, or joint disease
* History of asthma
* History of anaphylaxis
* Known history of intolerance to any formulation of intravenous iron

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Biomarkers of iron stores | 60 minutes
  Plantar flexion exercise as determined with a novel dynamic phosphorus magnetic resonance spectroscopy and imaging technique (31P-MRS & MRI) in heart failure patients (n=10) with and without functional iron deficiency. A spectrally selective three-dimensional turbo spin echo (3D-TSE) echo (3D-TSE) protocol for measurement of phosphocreatine recovery kinetics on a 3T Siemens MRI scanner as previously described (Siemens Medical Solutions, Erlangen, Germany).
Skeletal muscle bioenergetics using 31P- MRS Spectroscopy | 120 Minutes
  Plantar flexion exercise with 31P-MRS and MRI in heart failure patients (n=5) with functional iron deficiency. A spectrally selective three-dimensional turbo spin echo (3D-TSE) protocol for measurement of phosphocreatine recovery kinetics on a 3T Siemens MRI scanner (Siemens Medical Solutions, Erlangen, Germany).
  protocol for measurement of phosphocreatine recovery kinetics on a 3T Siemens MRI scanner as previously described (Siemens Medical Solutions, Erlangen, Germany).

SECONDARY OUTCOMES:
Functional Capacity | Six Minutes
  Subjects will be asked to walk along a 30 meter marked path in a corridor at a self-selected pace. Subjects will receive standardized instruction before and during the walking test. The distance walked after 6 minutes (meters) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Katz, MD, Principal Investigator — NYU Langone Health